CLINICAL TRIAL: NCT06621862
Title: Clinical Findings and Albuminuria as Predictors of Acute Kidney Injury in Patients With Acute Heart Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Hagar Mahmoud Hammad (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Hagar Mahmoud Hammad, Hagar Mahmoud Hammad, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AKI and heart failure
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure; Acute Kidney Injury; Albuminuria
Keywords: Heart failure; Acute Kidney Injury; Albuminuria
MeSH Terms: conditions — Heart Failure; Acute Kidney Injury; Albuminuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
assess the predictive value of clinical examination and proteinuria as early measures for acute kidney injury (AKI) in patient with acute heart failure and assessing their prognostic value as measures for mortality during hospital stay

DETAILED DESCRIPTION:
Heart failure (HF) is a chronic and progressive clinical syndrome induced by structural or functional cardiac abnormalities displaying either reduced (in HF with reduced ejection fraction (HFrEF)) or preserved (in HF with preserved ejection fraction (HFpEF)) left ventricular ejection fraction (LVEF) (1).

Current guidelines define the acute decompensated heart failure (ADHF) syndrome as the presence of new or worsening signs and symptoms of HF that often lead to hospitalization or an emergency department visit for intensification of therapies (2-4). Due to population growth and ageing, the total number of HF patients continues to rise. It is estimated that 64.3 million people live with HF worldwide. In developed countries, the prevalence of known HF is generally estimated at 1-2% of the general adult population.(3, 5)

Acute kidney injury (AKI) is a frequently occurring complication of critical illness, with severe impact on morbidity and mortality. Many studies focus on advanced measures, such as biomarkers or imaging for predicting AKI. These techniques are frequently time-consuming, costly, and are not available on a global scale. In contrast, variables obtained by clinical examination are readily available without limitations by set- tings or costs. Clinical examination signs and symptoms may reflect the underlying disease state and could therefore potentially be used to identify patients at risk for AKI . In addition, a few studies have specifically focused on the role of albuminuria in predicting adverse outcomes in heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients of 18 years and older who will be admitted to the ICU with acute heart failure (acute heart failure is defined according ESC guidelines 2021 which include Heart Failure with Reduced Ejection Fraction (HFrEF) EF <40% . Mid-Range Ejection Fraction (HFmrEF)(41 -46 %) , Preserved Ejection Fraction (HFpEF) EF ≥ 50%.

Exclusion Criteria:

* patients under the age of 18.

Patients with known chronic kidney disease (CKD) before ICU admission (CKD is defined as the presence of kidney damage or an estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73 mt2, persisting for 3 months or more, and or albuminuria more than 3.5 mg/mmol (12)

severe UTI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients of 18 years and older who will be admitted to the ICU with acute heart failure in Assiut University
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Assess the predictive value of clinical examination findings as and albuminuria for AKI in ADHF patients. | Baseline

SECONDARY OUTCOMES:
Assess effect of heart failure on the level of albuminuria | Baseline

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Levin A, Ahmed SB, Carrero JJ, Foster B, Francis A, Hall RK, Herrington WG, Hill G, Inker LA, Kazancioglu R, Lamb E, Lin P, Madero M, McIntyre N, Morrow K, Roberts G, Sabanayagam D, Schaeffner E, Shlipak M, Shroff R, Tangri N, Thanachayanont T, Ulasi I, Wong G, Yang CW, Zhang L, Robinson KA, Wilson L, Wilson RF, Kasiske BL, Cheung M, Earley A, Stevens PE. Executive summary of the KDIGO 2024 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease: known knowns and known unknowns. Kidney Int. 2024 Apr;105(4):684-701. doi: 10.1016/j.kint.2023.10.016. PMID 38519239
- [Result] Masson S, Latini R, Milani V, Moretti L, Rossi MG, Carbonieri E, Frisinghelli A, Minneci C, Valisi M, Maggioni AP, Marchioli R, Tognoni G, Tavazzi L; GISSI-HF Investigators. Prevalence and prognostic value of elevated urinary albumin excretion in patients with chronic heart failure: data from the GISSI-Heart Failure trial. Circ Heart Fail. 2010 Jan;3(1):65-72. doi: 10.1161/CIRCHEARTFAILURE.109.881805. Epub 2009 Oct 22. PMID 19850697
- [Result] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL. 2013 ACCF/AHA guideline for the management of heart failure: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):1810-52. doi: 10.1161/CIR.0b013e31829e8807. Epub 2013 Jun 5. No abstract available. PMID 23741057
- [Result] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Result] Hollenberg SM, Warner Stevenson L, Ahmad T, Amin VJ, Bozkurt B, Butler J, Davis LL, Drazner MH, Kirkpatrick JN, Peterson PN, Reed BN, Roy CL, Storrow AB. 2019 ACC Expert Consensus Decision Pathway on Risk Assessment, Management, and Clinical Trajectory of Patients Hospitalized With Heart Failure: A Report of the American College of Cardiology Solution Set Oversight Committee. J Am Coll Cardiol. 2019 Oct 15;74(15):1966-2011. doi: 10.1016/j.jacc.2019.08.001. Epub 2019 Sep 13. No abstract available. PMID 31526538
- [Result] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819